CLINICAL TRIAL: NCT00863902
Title: Single Dose Two-Way Crossover Fed Bioequivalence Study of Cetirizine Hydrochloride 10 mg Tablets in Healthy Volunteers
Brief Title: A Relative Bioavailability Study of Cetirizine HCl 10 mg Tablets Under Non-fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AAI-US-431
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-08-16 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Cetirizine; Healthy subjects
MeSH Terms: interventions — Cetirizine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cetirizine Hydrochloride (Experimental): Cetirizine Hydrochloride 10 mg tablets, single dose
  Interventions: Drug: Cetirizine Hydrochloride 10 mg tablets, single dose
- Zyrtec (Active Comparator): Zyrtec® 10 mg tablets, single dose
  Interventions: Drug: Zyrtec® 10 mg tablets, single dose

INTERVENTIONS:
Drug: Cetirizine Hydrochloride 10 mg tablets, single dose — A: Experimental Subjects received Shasun Chemicals and Drugs Ltd. formulated products under fed conditions
  Other Names: Cetirizine
  Arms: Cetirizine Hydrochloride
Drug: Zyrtec® 10 mg tablets, single dose — B: Active comparator Subjects received Pfizer Inc. formulated products under fed conditions
  Other Names: Cetirizine
  Arms: Zyrtec

SUMMARY:
To determine the pharmacokinetics and bioequivalence of cetirizine hydrochloride formulations after administration of single doses to normal healthy subjects under fed conditions. These data were to be evaluated statistically to determine if the products meet bioequivalence criteria.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Single-dose two-way, crossover bioequivalence study with an adequate washout period (7 days) between the two periods of the study and with an equal number of subjects randomly assigned to receive the study test (Treatment A) and study reference (Treatment B).

Official Title: Single Dose Two-Way Crossover Fed Bioequivalence Study of Cetirizine Hydrochloride 10 mg Tablets in Healthy Volunteers

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects at least 18 years of age.
2. Informed of the nature of the study and provide their written informed consent.
3. Have a body mass index2 between 18 and 30 and weighing at least 110 pound.
4. In good health as determined by lack of clinically significant abnormalities in health assessments performed at screening as judged by the physician.

Exclusion Criteria:

1. Hypersensitivity to cetirizine hydrochloride (Zyrtec®) or related compounds.
2. Conditions that affect the absorption, metabolism or passage of drugs out of the body, e.g., sprue, celiac disease, Crohn's disease, colitis, liver, kidney or thyroid conditions.
3. Recent history (within 1 year) of mental illness, drug addiction, drug abuse or alcoholism.
4. A hematocrit value of ≤ 33.0 % for females and ≤ 37.0 % for males.
5. Donation of greater than 500 ml of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.
6. Received an investigational drug within the 4 weeks prior to study dosing.
7. Currently taking any systemic prescription medications, except for oral/cutaneous/vaginal hormone contraceptives, within the 7 days prior to study dosing or over-the-counter medication within 3 days of study dosing. This prohibition does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physician. Any nonprescription medication consumption reported will be reviewed by the investigator prior to dosing. At the discretion of the investigator these volunteers may be enrolled if the medication is not anticipated to alter study integrity.
8. Regular smoking of more than 5 cigarettes weekly or the regular daily use of nicotine-containing products beginning 3 months before study medication administration through the final evaluation.
9. If female, the subject is lactating or has a positive pregnancy test at screening and prior to each of the treatment periods. Females must use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or her partner are: oral contraceptives/patches, progestin injection or implants, condom with spermicide, diaphragm with spermicide, IUD, vaginal spermicidal or hormonal suppository, surgical sterilization of themselves or their partner(s) or abstinence. Females taking oral contraceptives/patches must have taken them consistently for at least three months prior to receiving study medication.
10. Grapefruit beverages or foods beginning 7 days before each study medication administration and alcohol, caffeine or xanthine beverages or foods beginning 24 hours before each study medication administration through the last PK sample of each period. Such restricted items include coffee, tea, iced tea, Coke®, Pepsi®, Mountain DeW®, chocolate, brownies, etc.
11. Regular use of any drugs known to induce or inhibit hepatic drug metabolism (examples include barbiturates, carbamazepine, rifampin, phenylhydantoins, phenothiazines, cimetidine,omeprazole, macrolides, imidazoles, fluoroquinolones) within 30 days prior to study administration.
12. Positive test results for: HIV, Hepatitis B surface antigen, Hepatitis C antibody at screening.
13. Positive test results for: drugs of abuse or pregnancy at screening and prior to each dosing period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2006-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Evin H. Sides III,, MD, Principal Investigator — AAI Clinic (AAIPharma Inc.)
Locations (1):
- AAIPharma Inc.- AAI Clinic, Morrisville, North Carolina, United States